CLINICAL TRIAL: NCT04758650
Title: Phase II Study to Evaluate the Clinical Potential of 68GaNOTA-Anti-MMR-VHH2 for in Vivo Imaging of MMR-expressing Macrophages by Means of Positron Emission Tomography (PET) in Oncological Lesions,Cardiovascular Atherosclerosis,Syndrome With Abnormal Immune Activation and sarcoïdosis
Brief Title: Study of 68GaNOTA-Anti-MMR-VHH2 in Oncological Lesions, Cardiovascular Atherosclerosis, Syndrome With Abnormal Immune Activation and sarcoïdosis
Acronym: MITRAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UZBRU_VHH2_2; 2020-002483-31 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Solid Malignancy Located in the Head and Neck; Cancer; Carotid Stenosis; Atherosclerosis of Artery; Hodgkin Lymphoma, Adult; Non Hodgkin Lymphoma; HLH; Cardiac Sarcoidosis; Sarcoidosis
MeSH Terms: conditions — Neoplasms; Carotid Stenosis; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sarcoidosis

STUDY DESIGN:
Intervention Model Description: The trial consists of 7 different patient cohorts that are each investigated using a new diagnostic imaging radiopharmaceutical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer, lymphoma, carotid plaque, patients suspected for HLH, sarcoidosis (Experimental): Cohort 1: Patients diagnosed with pathology malignancies of the head and neck
  Cohort 2: Patients diagnosed with any malignancy with a solid component
  Cohort 3: Patients diagnosed with carotid plaque, planned for SOC carotid endarterectomy
  Cohort 4: Patients with a biopsy-proven Hodgkin or non-Hodgkin lymphoma
  Cohort 5: Patients suspected for HLH, planned for (SOC) bone marrow in case it is not done before
  Cohort 6 : Patients with endomyocardial biopsy proven or suspected cardiac sarcoïdosis
  Cohort 7 : Patients with biopsy-proven sarcoïdosis
  Interventions: Drug: 68GaNOTA-Anti-MMR-VHH2

INTERVENTIONS:
Drug: 68GaNOTA-Anti-MMR-VHH2 — All subjects will receive at least one single intravenous injection of the IMP followed by a total body PET/CT prior to receiving standard-of-care therapy.
  For patients in cohorts 1 and 2 : an optional injection of the IMP during or after therapy can be administered if a patient is treated with non-surgical modalities. Patients in cohorts 6 and 7 who receive standard-of-care treatment can receive an optional injection of the IMP.
  Other Names: MMR-PET/CT

SUMMARY:
Phase II study to evaluate the clinical potential of 68GaNOTA-anti-MMR-VHH2 for in vivo imaging of Macrophage Mannose Receptor (MMR)-expressing Macrophages by means of Positron Emission Tomography (PET) in patients with oncological lesions in need of non-surgical therapy, patients with cardiovascular atherosclerosis, syndrome with abnormal immune activation and sarcoïdosis.

ELIGIBILITY:
COHORT SPECIFIC INCLUSION CRITERIA:

* COHORT 1:

  - Patients who have given informed consent

  - Patients at least 18 years old

  - Patients with : A) biopsy-proven solid malignancy located in the head and neck, independent of tumour stage or pathological subtype, or B) suspected malignancy in the head and neck, planned for biopsy
  * In order to minimize partial volume effect, the diameter of at least 1 tumour lesion should be ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions.
  * Patients who already participated in the trial and who are diagnosed with progressive or recurrent disease can be re-included if all inclusion criteria and none of the exclusion criteria apply.
* COHORT 2:

  * Patients who have given informed consent
  * Patients at least 18 years old
  * Patient with a biopsy proven local, locally advanced or metastatic malignancy with a solid component that is at least ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions.
  * The patient is planned for immune checkpoint inhibition treatment, either or not combined with other systemic therapies.
  * Patients who already participated in the trial and who are diagnosed with progressive or recurrent disease can be re-included if all inclusion criteria and none of the exclusion criteria apply
* COHORT 3:

  * Patients who have given informed consent
  * Patients at least 18 years old
  * Patients planned for the surgical removal of an atherosclerotic plaque of the carotid artery, consisting of endarterectomy.
* COHORT 4:

  * Patients who have given informed consent
  * Patients at least 18 years old
  * Patient with a biopsy-proven Hodgkin or non-Hodgkin lymphoma
  * At time of inclusion, the patient presents with at least 1 lymphoma lesion of which the diameter should be ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions.
  * Diagnostic tissue sample is available for immunohistochemistry analysis, that was obtained < 3 months prior to patient inclusion.
  * 18F-FDG-PET/CT has been performed < 3 months prior to patient inclusion
  * The patients are eligible for systemic treatment, radiotherapy or a combination of both.
* COHORT 5:

  * Patients who have given informed consent
  * Patients at least 18 years old
  * Patients with suspicion of HLH, based on either a previous bone marrow sample showing hemofagocytis or based on the presence of at least 3 risk criteria as follows :
  * Fever ≥ 38,5°C
  * Splenomegaly
  * Bicytopenia, with at least 2 of the 3 following parameters:
  * Hb < 9 g/dl and/or
  * Platelets < 100 000/ml and/or
  * Neutrophils < 1000/ml
  * Hypertriglyceridemia (fasting > 265 mg/dl)µ
  * Ferritin > 500 ng/ml
* COHORT 6:

  * Patients who have given informed consent
  * Patients at least 18 years old
  * Patients with :

A) Endomyocardial biopsy-proven cardiac sarcoidosis (CS) or B) suspected cardiac sarcoidosis based on the 2014 Hearth Rythm Society Expert Consensus Statement on the Diagnosis and Management of Arrhytmias Associated with Cardiac Sarcoidosis. At least one of the following criteria should be met :

* Steroid +/- Immunosuppressant responsive cardiomyopathy or heart block
* Unexplained reduced left ventricular ejection fraction (LVEF) <40%
* Unexplained sustained (spontaneous or induced) ventricular tachycardia (VT)
* Mobitz type II 2nd-degree heart block or 3rd-degree heart block
* Patchy uptake on dedicated cardiac PET (in a pattern consistent with CS)
* Late Gadolinium Enhancement on Cardiovascular Magnetic Resonance (in a pattern consistent with CS)
* Positive gallium uptake (in a pattern consistent with CS)
* Histological Diagnosis from Myocardial Tissue
* Patients already included in cohort 7 with progression to cardiac sarcoidosis

  *COHORT 7:
* Patients who have given informed consent
* Patients at least 18 years old
* Patients with biopsy-proven sarcoidosis

GENERAL EXCLUSION CRITERIA:

* Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher.
* Pregnant patients.
* Breast feeding patients.
* Patients with any serious active infection.
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test radiopharmaceutical.
* Patients who cannot communicate reliably with the investigator.
* Patients who are unlikely to cooperate with the requirements of the study.
* Patients who are unwilling and/or unable to give informed consent.
* Patients at increased risk of death from a pre-existing concurrent illness.
* When a patient exhibits symptoms correlated with SARS-CoV-2, the patient should be tested using the standard of care testing protocol, prior to inclusion. When the test results indicate an active SARS-CoV-2-infection, the patient is excluded for this trial.

COHORT SPECIFIC EXCLUSION CRITERIA

* COHORT 2

  * Patients with a biopsy-proven Hodgkin or non-Hodgkin lymphoma
  * Patients diagnosed with any malignancy of the head and neck. These patients can be included into Cohort I.
* COHORT 7 - Patients eligible for cohort 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-01-26 (Estimated)

PRIMARY OUTCOMES:
Correlation of IMP uptake before start of treatment in malignant lesions of the head and neck with either treatment response during or after radiotherapy or systemic treatment, or with immunohistological MMR-staining in patients with surgical treatment | up to 5 years
  Uptake will be measured in cancer lesions on PET/CT 1. Treatment response will be evaluated by assessing time to treatment failure and by assessment of status of patients for treatment failure (Y/N) at 6 and 12 months after start of treatment or immunological MMR staining
Correlation of uptake of 68GaNOTA-Anti-MMR-VHH2 before start of treatment in solid cancer lesions with time to treatment failure after systemic treatment with immune checkpoint inhibition, either or not combined with other systemic therapies. (cohort 2) | up to 5 years
  Uptake will be measured in cancer lesions on PET/CT 1. Treatment response will be evaluated by assessing time to treatment failure and by assessment of status of patients for treatment failure (Y/N) at 6 months and 12 months after start of treatment
Correlation of uptake of 68GaNOTA-Anti-MMR-VHH2 in atherosclerotic carotid plaques before surgery with the immunohistological MMR-staining of the excised atherosclerotic carotid plaque.(cohort 3) | Resection of lesion up to 21 days after PET/CT
  Uptake in excised atherosclerotic plaque on PET/CT 1. Immunohistological MMR staining of excised atherosclerotic plaque, scored visually by interpreter
Correlation of uptake of 68GaNOTA-Anti-MMR-VHH2 in lymphoma-related lesions before start of treatment in Hodgkin and non-Hodgkin lymphoma patients (cohort 4). | up to 5 years
  Uptake will be measured in lymphoma-related lesions on MMR-PET/CT 1
Correlation of uptake of 68GaNOTA-Anti-MMR-VHH2 in central bone on PET/CT with the presence of hemophagocytosis in bone marrow samples, and the presence of clinical risk factors (cohort 5). | up to 5 years
  Uptake in bone marrow on MMR-PET/CT 1. Bone marrow aspirate or trephine biopsy, scored individually by interpreter. Results of additional blood sample analysis to determine clinical risk factor
To investigate the uptake of 68GaNOTA-Anti-MMR-VHH2 in cardiac sarcoidosis on PET/CT in patients with endomyocardial biopsy proven or suspected cardiac sarcoidosis (cohort 6) | up to 5 years
  Uptake in lesions with known or suspected cardiac sarcoidosis on MMR-PET/CT on PET/CT1
To investigate the uptake of 68GaNOTA-Anti-MMR-VHH2 in sarcoidosis on PET/CT in patients with biopsy-proven sarcoidosis (cohort 7) | up to 5 years
  Uptake in lesions involved with sarcoidosis on MMR-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lahoutte, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Uz Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No